## **CCB-01**

## STUDY PROTOCOL

A Phase 1b/2a open-label, multi-center study to assess the safety, efficacy and pharmacokinetics of intrapatient dose-adjusted brequinar and inhibition of dihydroorotate dehydrogenase (DHODH) in adult subjects with acute myelogenous leukemia (AML)

NCT03760666

Statistical Analysis Plan – 09/11/2019



# Sponsor Approval Form

| Date Tit Sep 2019 Protocol: CCB-01 | Project: | YYA36071 | Sponsor: | Clear Cr | eek Bio, Inc. |
|---|---|---|---|---|---|
| Telemann File name (for electronic documents) | Date: | 11 Sep 2019 | Protocol: | CCB-01 | |
| □ * System Configuration □ * Rights and Roles □ * eCRF Design – PDF of forms □ * Edit Check Specifications □ eRF Completion Guidelines □ SAE Reconciliation Guidelines □ Coding Report □ Randomization Schedule Specification □ Unblinding Plan □ Study Data Transfer □ Site Payment Criteria Specifications □ SDTM Transfer □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ 20190911 CCB-01 YYA36071 SAP v1.0.doc □ Statistical Analysis Plan – data display shells □ Statistical Report/Summary □ Other, specify: □ Statistical Report/Summary □ Other, specify: □ Statistical Report Summary □ Other, specify: □ Statistical Report Summary □ Other, specify: □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: ALKA Ahuja [Sponsor Title]; [Sponsor Company] 11 September 2019 | | and distribution of the state o | | | |
| □ * System Configuration □ * Rights and Roles □ * eCRF Design – PDF of forms □ * eCRF Completion Guidelines □ * ECRF Completion Guidelines □ * Configuration Schedule Specification □ Randomization Schedule Specification □ Randomization Plan □ Unblinding Plan □ Study Data Transfer Requirements □ SDTM Specifications □ CDF Specifications □ CDF Specifications □ Step Payment Criteria Specifications □ Statistical Analysis Plan – text □ 20180911 CCB-01 YYA36071 SAP v1.0.doc □ Statistical Analysis Plan – text □ 20190911 CCB-01 YYA36071 TLF Shells.doc □ Statistical Reporting – TLF Delivery □ Statistical Report Summary □ Other, specify: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: ALKA Ahuja [Sponsor Title]; [Sponsor Company] 11 September 2019 | Item(s) Sub | mitted for Approval | File | name (for | electronic documents) |
| □ *Rights and Roles □ *eGRF Design – PDF of forms □ *Edit Check Specifications □ eCRF Completion Guidelines □ SAE Reconciliation Guidelines □ Coding Report □ Randomization Schedule Specification □ Unblinding Plan □ Unblinding Plan □ Unblinding Plan □ Study Data Transfer Requirements □ SDTM Specifications □ SDTM Transfer □ CDF Specifications □ SDTM Transfer □ CDF Specifications □ SDTM Transfer □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Report/Summary □ Statistical Report/Summary □ Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: ALKA Ahuja [Biostatistician]; Novella Clinical □ [Sponsor Title]; [Sponsor Company] 11 September 2019 | the state of the s | | | | |
| □ * eCRF Design – PDF of forms □ * Edit Check Specifications □ eCRF Completion Guidelines □ Coding Report □ Randomization Schedule Specification □ Randomization Schedule Specification □ Randomization Plan □ Unblinding Plan □ Study Data Transfer Requirements □ SDTM Specifications □ SDTM Specifications □ SDTM Specifications □ SDTM Transfer □ CDF Specifications □ Site Payment Criteria Specifications □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Reporting – TLF Delivery □ Statistical Repor | | | | | |
| □ *Edit Check Specifications □ cRF Completion Guidelines □ SAE Reconciliation Guidelines □ SAE Reconciliation Guidelines □ Coding Report □ Randomization Schedule Specification □ Randomization Plan □ Unblinding Plan □ Unblinding Plan □ Study Data Transfer Requirements □ SDTM Specifications □ SDTM Transfer □ CDF Specifications □ SDTM Transfer □ CDF Specifications □ Site Payment Criteria Specifications □ Statistical Analysis Plan - text □ Statistical Analysis Plan - text □ Statistical Analysis Plan - 20190911 CCB-01 YYA36071 SAP v1.0.doc □ Statistical Analysis Plan - data display shells □ Statistical Reportifyammary □ Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | | | | | |
| GCRF Completion Guidelines SAE Reconciliation Guidelines Coding Report Randomization Schedule Specification Randomization Plan Unblinding Plan Study Data Transfer Requirements SDTM Specifications SDTM Transfer CDF Specifications CDF Specifications CDF Specifications Stitustical Analysis Plan − text Statistical Analysis Plan − text Statistical Analysis Plan − text Statistical Reportifyammary Statistical Reportifyammary Statistical Reportifyammary Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Movella Clinical performs QC and documents successful implementation of changes. (Standard practice) naddition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) | | | | 4.1 | |
| □ SAE Reconciliation Guidelines □ Coding Report □ Randomization Schedule Specification □ Randomization Plan □ Unbilinding Plan □ Unbilinding Plan □ Study Data Transfer Requirements □ SDTM Specifications □ CDF Specifications □ CDF Test Transfer □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Reporting – TLF Delivery □ Statistical Report/Summary □ Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: ALRA ANUJA Alka Ahuja [Biostatistician]; Novella Clinical 11 September 2019 | | | | | |
| Randomization Schedule Specification Randomization Plan Unblinding Plan Study Data Transfer Requirements SDTM Specifications SDTM Specifications ODF Specifications ODF Test Transfer Site Payment Criteria Specifications Statistical Analysis Plan – text 20190911 CCB-01 YYA36071 SAP v1.0.doc Statistical Analysis Plan – data display shells Statistical Reporting – TLF Delivery Statistical Report/Summary Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: Nonel *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: ALRA Ahuja Rika Ahuja Rika Ahuja Rika Ahuja Risponsor Taite]; (Sponsor Company) 11 September 2019 | | | | | |
| □ Randomization Plan □ Inbilinding Plan □ Study Data Transfer Requirements □ SDTM Specifications □ SDTM Transfer □ CDF Specifications □ SDTM Transfer □ CDF Specifications □ SDTM Transfer □ Site Payment Criteria Specifications ☑ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Report/summary □ Statistical Report/summary □ Other, specify: □ Other, specify: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: ALRA Ahuja Biostatistician]; Novella Clinical □ Isponsor Title]; [Sponsor Company] 11 September 2019 | ☐ Coding R | eport | | | |
| □ Study Data Transfer Requirements □ SDTM Specifications □ SDTM Transfer □ CDF Specifications □ CDF Test Transfer □ Steatistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – data display shells □ Statistical Reporting – TLF Delivery □ Statistical Reporting – TLF Delivery □ Statistical Report/Summary □ Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: ALRA Ahuja Alka Ahuja Alka Ahuja [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | Randomiz | ration Schedule Specification | | | |
| Study Data Transfer Requirements □ SDTM Specifications □ CDF Specifications □ CDF Specifications □ CDF Test Transfer □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Reporting – TLF Delivery □ Statistical Reporting – Text | Randomiz | zation Plan | | | |
| □ SDTM Specifications □ SDTM Transfer □ CDF Specifications □ CDF Test Transfer □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Reporting – TLF Delivery □ Statistical Reporting – TLF Delivery □ Statistical Report/Summary □ Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: ALRA ANUJA Alka Ahuja [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | Unblindin | g Plan | | | |
| □ SDTM Transfer □ CDF Test Transfer □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – 20190911 CCB-01 YYA36071 SAP v1.0.doc □ Statistical Reporting – TLF Delivery □ Statistical Report/Summary □ Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Company] 11 September 2019 | ☐ Study Dat | ta Transfer Requirements | | | |
| □ CDF Specifications □ CDF Test Transfer □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ Statistical Analysis Plan – text □ Statistical Analysis Plan – data display shells □ Statistical Report/Summary □ Statistical Report/Summary □ Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | ☐ SDTM Sp | ecifications | | | |
| □ CDF Test Transfer □ Site Payment Criteria Specifications □ Statistical Analysis Plan – text □ Statistical Analysis Plan – 20190911 CCB-01 YYA36071 SAP v1.0.doc □ Statistical Analysis Plan – 20190911 CCB-01 YYA36071 TLF Shells.doc □ data display shells □ Statistical Reporting – TLF Delivery □ Statistical Report/Summary □ Other, specify: □ Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: ■ [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Biostatistician]; Novella Clinical [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | SDTM Tra | ansfer | | | |
| Site Payment Criteria Specifications Statistical Analysis Plan – text Statistical Analysis Plan – data display shells Statistical Analysis Plan – data display shells Statistical Report/Summary Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | ☐ CDF Spe | cifications | | | |
| Statistical Analysis Plan – text Statistical Analysis Plan — data display shells Statistical Reporting – TLF Delivery Statistical Report/Summary Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | CDF Test | Transfer | | | |
| Statistical Analysis Plan − data display shells Statistical Reporting – TLF Delivery Statistical Report/Summary Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | | | | | |
| data display shells Statistical Reporting – TLF Delivery Statistical Report/Summary Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Company] 11 September 2019 | | | 201 | 90911 CCI | 3-01 YYA36071 SAP v1.0.doc |
| Statistical Reporting – TLF Delivery Statistical Report/Summary Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja Biostatistician]; Novella Clinical Sponsor Name] Sponsor Company] 11 September 2019 | | | 201 | 90911 CCI | 3-01 YYA36071 TLF Shells.doc |
| □ Statistical Report/Summary □ Other, specify: Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: □ Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) □ In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: □ With proof of changes (i.e. screen shots or annotated PDFs). □ With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Biostatistician]; Novella Clinical [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | I control to the second | | | | |
| Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Company] 11 September 2019 | | | | | |
| Signature indicates sponsor approved as delivered, unless modifications are listed/referenced below: • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Company] 11 September 2019 | | | | | |
| • [None] *For approvals of documents with changes post-production, please select one of the following methods to verify that the changes have been completed successfully: Novella Clinical performs QC and documents successful implementation of changes. (Standard practice) In addition to Novella Clinical QC, Sponsor will verify changes before changes are implemented in production: With proof of changes (i.e. screen shots or annotated PDFs). With User Acceptance Testing (UAT) (May affect timeline and/or cost) Signatures: Alka Ahuja [Sponsor Name] [Sponsor Title]; [Sponsor Company] 11 September 2019 | Other, sp | ecify: | | | |
| Alka Ahuja [Biostatistician]; Novella Clinical 11 September 2019 Ballara Powers [Sponsor Name] [Sponsor Title]; [Sponsor Company] 23 Sept 2019 | *For approva<br>changes hav<br>Nov<br>In a<br>pro | [None] als of documents with change we been completed successful wella Clinical performs QC an addition to Novella Clinical QC duction: With proof of changes (i.e. so | es <u>post-prod</u><br>illy:<br>d documen<br>C, Sponsor<br>creen shots | duction, pleats success will verify or annotate | ease select one of the following methods to verify that the sful implementation of changes. (Standard practice) changes before changes are implemented in ted PDFs). |
| Alka Ahuja [Biostatistician]; Novella Clinical 11 September 2019 [Sponsor Name] [Sponsor Title]; [Sponsor Company] 23 Sept 2019 | Signatures | s: | | | |
| [Biostatistician]; Novella Clinical [Sponsor Title]; [Sponsor Company] 11 September 2019 | | V | | | Barbara Powers |
| 11 September 2019 23 Sept 2019 | | | | | |
| Deta | [Biostatistic | cianj; Novelia Clinical | | 1 | |
| Data | 11 Septem | ber 2019 | | 1 | 23 Sept 2019 |
| | | | | 1 | Date |

Novella may make necessary corrections to spellings, punctuation, and obvious errors without further approval of the Sponsor.

Document Number: NVA\_FM\_DO189 Revision 13 Effective Date: 04Oct2016
DCN #1484 Document Title: Sponsor Approval Form Page 1 of 1

# Clear Creek Bio, Inc. Protocol #: CCB-01

A Phase 1b/2a open-label, multi-center study to assess the safety, efficacy and pharmacokinetics of intrapatient dose-adjusted brequinar and inhibition of dihydroorotate dehydrogenase (DHODH) in adult subjects with acute myelogenous leukemia (AML)

## **Statistical Analysis Plan**

#### Version 1.0

Document last saved: 18-Jan-2022 9:43 AM

Prepared for:

Clear Creek Bio, Inc. 585 Massachusetts Avenue, 4<sup>th</sup> Floor Cambridge, MA 02139 USA Prepared by:

IQVIA Biotech 1700 Perimeter Park Dr. Morrisville, NC 27560 USA

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372 Document Title: Statistical Analysis Plan Template P a g e | i

## **Statistical Analysis Plan Signatures**

| Prepared by: | Alka Ahuja, MS IQVIA Biotech 1700 Perimeter Park Drive Morrisville, NC 27560 USA Tel: +1 919-336-9323 Fax: +1 919-484-7727 alka.ahuja@iqvia.com | |
|---|---|---|
| Approved by: | | |
| | D 1 D MCN DID | |
| | Barbara Powers, MSN, PhD<br>Clinical Development, Clear Creek Bio, Inc. | Date |
| | Alka Ahuja, MS | Date |
| | Biostatistician II, IQIVA Biotech | |

Effective Date: 13-Apr-2015 Page | ii Document Number: FORM 694.01 Document Title: Statistical Analysis Plan Template DCN # 1372

## **Table of Contents**

| Statistical Analysis Plan Signatures | ii |
|---------------------------------------------------------|-----|
| Table of Contents | iii |
| List of Abbreviations | v |
| I.Introduction | 1 |
| II.Protocol Objectives | 1 |
| A. Primary | 1 |
| B. Secondary | 1 |
| C. Exploratory | |
| III.Study Endpoints | |
| A. Primary Endpoints | |
| B. Secondary Endpoints C. Exploratory Endpoints | |
| IV.Study Design | |
| A. Design Overview B. Study Population | |
| C. Sample Size Predictions | |
| V.General Analytical Considerations | |
| A. Data Sources | |
| B. Multiple Study Centers | |
| C. Definition of Baseline | |
| D. Missing Data | |
| E. Analysis Populations F. Data Display Characteristics | |
| VI.Subject Accountability | |
| • | |
| A. Analysis Populations B. Disposition | |
| C. Subject Characteristics | |
| D. Protocol Deviations | |
| VII.Safety Analyses | 9 |
| A. Exposure | 9 |
| B. DHO Plasma Levels | 10 |
| C. Dose Limiting Toxicities | |
| D. Adverse Events E. Deaths | |
| F. Clinical Laboratory Results | |
| G. Vital Signs | |
| H. 12-Lead Electrocardiogram | |
| I FCOG Performance Status | 12 |

### Clear Creek Bio, Inc. / Protocol: CCB-01 IQVIA Biotech (Confidential) Project # YYA36071

| J. | Physical Examination | 12 |
|------------|--------------------------------------|----|
| K. | Concomitant Medications | 12 |
| L. | Blood Transfusions | 13 |
| VIII.Effic | acy Analyses | 13 |
| A. | Disease Response | 13 |
| B. | Clinical Benefit | 14 |
| IX.Pharma | acokinetic Analyses | 14 |
| X.Explora | ntory Analyses | 15 |
| XI.Chang | es from Analyses Planned in Protocol | 16 |
| XII.Refere | ences | 17 |

## **List of Abbreviations**

| A11 | D. 6'' 11' |
|---|---|
| Abbreviation | Definition |
| ANC | Absolute neutrophil count |
| AE | Adverse event |
| AML | Acute myelogenous leukemia |
| $\mathrm{AUC}_{0	ext{-last}}$ | Area under curve from time 0 to time of last measurable |
| | concentration. |
| $\mathrm{AUC}_{0	ext{-inf}}$ | Area under curve from time 0 to infinity |
| BOR | Best overall response |
| BSA | Body surface area |
| CI | Confidence interval |
| CL | Systemic clearance |
| $C_{max}$ | Maximum observed plasma concentration |
| CR | Complete remission |
| CRh | CR with partial hematological recovery |
| Cri | CR with incomplete hematological recovery |
| $C_{ss}$ | Observed concentration at steady state |
| CTCAE | Common terminology criteria for adverse events |
| DHO | Dihydroorotate |
| DHODH | Dihydroorotate dehydrogenase |
| DLT | Dose-limiting toxicity |
| DNA | Deoxyribonucleic acid |
| DOR | Duration of response |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic case report form |
| EFS | Event-free survival |
| FISH | Fluorescence in situ hybridization |
| Hgb | Hemoglobin |
| mg | Milligram |
| $m^2$ | Meters squared |
| MedDRA | Medical dictionary for regulatory affairs |
| MLFS | Morphologic leukemia-free state |
| NCI CTCAE | National Cancer Institute Common Terminology Criteria |
| | for Adverse Events |
| ORR | Overall response rate |
| OS | Overall survival |
| PK | Pharmacokinetic(s) |
| PR | Partial remission |
| PT | Preferred term |
| SAP | Statistical analysis plan |
| SI units | International system of units |
| SOC | System organ class |
| $t_{1/2}$ | Elimination half-life |
| $T_{max}$ | Time to maximum plasma concentration |
| TEAE | Treatment-emergent adverse event |
| TI | Transfusion independence |
| TLF | Tables, listings, and figures |

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372 Document Title: Statistical Analysis Plan Template Effective Date: 13-Apr-2015

Clear Creek Bio, Inc. / Protocol: CCB-01 IQVIA Biotech (Confidential) Project # YYA36071

 $V_{ss}$  Volume of distribution at steady state WHODD World health organization drug dictionary

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372 Document Title: Statistical Analysis Plan Template Effective Date: 13-Apr-2015 P a g e | vi

#### I. Introduction

This Statistical Analysis Plan (SAP) presents details of the analyses required to address the study aims of protocol CCB-01 version 6.0, dated 30 April 2019. The study is a phase 1b/2a open-label, multi-center trial with a purpose to evaluate the safety, efficacy, and pharmacokinetics (PK) of the drug oral brequinar in subjects 18 years or older with relapsed/refractory acute myeloid leukemia (AML), as well as to determine the inhibitory level of brequinar in blocking the enzyme "dihydroorotate dehydrogenase" (DHODH).

Safety and tolerability of brequinar will be assessed via adverse event (AE) monitoring, clinical laboratory safety tests, physical examinations, vital signs measurements, 12-lead electrocardiogram (ECG) readings, and bone marrow sampling. Specific efficacy endpoints of disease response, and PK profiles of brequinar and dihydroorotate (DHO) plasma levels will also be characterized.

This SAP has been developed and approved prior to database lock and data analysis. All analyses will be conducted after clinical trial data are entered into the database, discrepancies resolved, and the database is authorized (closed to further changes). Any deviations from the SAP will be documented as such in the study report.

Production and quality control of statistical analyses and accompanying tables, listings, and figures (TLFs) will be the responsibility of IQVIA Biotech located in Morrisville, North Carolina, United States.

#### II. **Protocol Objectives**

#### A. Primary

The protocol lists the following primary objective:

To determine the safety and tolerability of brequinar and the DHODH inhibitory activity of brequinar in adult subjects with AML.

#### **B.** Secondary

The protocol lists the following secondary objectives:

To determine the overall response rate (ORR) including complete remission (CR), CR with incomplete hematologic recovery (CRi), morphologic leukemia-free state (MLFS), partial remission (PR) (criteria as defined in the ELN Guidelines, by **Dohner et al.**, 2017) and complete remission with partial hematological recovery (CRh).

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372 

- To assess the rate of overall survival (OS) and event-free survival (EFS).
- To evaluate duration of response (DOR).
- To characterize the pharmacokinetic (PK) profile of brequinar.
- To characterize the DHO plasma levels after oral dosing with brequinar.

### C. Exploratory

The protocol lists the following exploratory objectives:

- To assess the relationship between DHODH inhibition and the efficacy and safety of brequinar.
- To evaluate molecular and cellular biomarkers that may be predictors of antitumor level and/or treatment resistance including cytogenetics, molecular profiling, and flow cytometry during and after treatment.
- To evaluate global gene expression profiles, deoxyribonucleic acid (DNA)methylation profiles, and other potential prognostic markers to explore predictors of antitumor activity and/or resistance to treatment.

#### III. **Study Endpoints**

### A. Primary Endpoints

The study protocol defines primary endpoints as safety/tolerability and DHO level relationship with safety and therapeutic brequinar levels.

Safety/tolerability, assessed at each study visit using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, will be evaluated for each subject as follows:

- Through Day 42, Grade 3 or higher, treatment-emergent, study drug-related, non-hematologic AE will be considered unacceptable toxicity with the following exceptions:

| Condition | Exception Description |
|---|---|
| Nausea/ Emesis | Grade 3 nausea and/or emesis resolving to less than or equal to Grade 2 |
| | or baseline within 1 week after the use of an optimal antiemetic regimen |
| | based on standard practice. |
| Diarrhea | Grade 3 diarrhea resolving to less than or equal to Grade 1 or baseline |
| | within 1 week after receiving the maximal supportive therapy based on |
| | standard practice. |
| Laboratory | Asymptomatic Grade 3 laboratory abnormalities that are not considered |
| abnormalities | to be clinically significant. |
| Mucositis | Grade 3 with duration < 1 week. |
| Fatigue | Grade 3 with duration < 2 weeks. |

Effective Date: 13-Apr-2015 Document Number: FORM 694.01 DCN # 1372 Document Title: Statistical Analysis Plan Template 

- After 42 days of treatment, criteria for unacceptable safety will be expanded to include hematologic AEs defined as:
  - Prolonged neutropenia with ANC < 500 from start of therapy in the absence of disease.
  - > Grade 4 neutropenia.
  - And/or > Grade 4 thrombocytopenia with a hypocellular bone marrow and no greater than 5% marrow blasts lasting for > 2 weeks.
- After 42 days of treatment, in expansion cohort subjects, the definition of unacceptable safety will include signs of hepatotoxicity (an episode of > Grade 2 toxicity for ALT and AST).

#### **Secondary Endpoints**

The following secondary endpoints will be analyzed:

- ORR including CR, CRi, CRh, MLFS, or PR.
- · Rates of OS and EFS.
- Duration of response.
- PK profile of brequinar.
- DHO plasma profile.

#### C. Exploratory Endpoints

The following endpoints will be explored:

- Relationship between DHODH inhibition and the efficacy and safety of brequinar.
- Antitumor level based on molecular and cellular biomarkers including cytogenetics, molecular profiling, and flow cytometry during and after treatment.
- Global gene expression profiles, DNA methylation profiles, and other potential prognostic markers to explore predictors of antitumor activity and/or resistance to treatment.

#### IV. **Study Design**

#### A. Design Overview

This will be a phase 1b/2a multi-center, open-label, non-randomized clinical trial to assess the safety, tolerability and efficacy of dose-adjusted brequinar in adult subjects with AML. The study will also assess the inhibition of DHODH and the PK profile of brequinar in plasma. Intra-subject dosing will be adjusted based on safety/tolerability, brequinar PK, and DHO levels.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372  Up to 27 subjects are planned to be entered in this trial. Cohort 1 was planned to have 6 subjects, but enrollment was stopped after 5 subjects when brequinar PK and DHO results became available. These results led to study design changes as described here. The sixth subject will not be enrolled in Cohort 1.

Cohort 2 will enroll approximately 6 subjects, followed by an expansion cohort of approximately 15 subjects. All subjects in Cohort 2 will start with a 500 mg/m<sup>2</sup> dose once-weekly. Brequinar PK and DHO samples will be obtained for these subjects in Week 1 and results used to make decisions about the Week 2 once-weekly dose. Brequinar PK and DHO samples will also be obtained for Week 2 and the results used to make decisions about Week 3 dose frequency (once or twice-weekly) and the dose. The dose will be adjusted for each subject to meet the twice-weekly brequinar PK and 72-hour DHO criteria, and the Week 2 procedures may be repeated if needed until the twice-weekly dose is found.

After both the brequinar PK and 72-hour DHO level meet criteria described in the Individual Dose Adjustment Guidelines as described in Protocol Section 8.5, a subject may move to twice-weekly dosing on a continuing basis as tolerated. The twice-weekly dose may be further adjusted using 84-hour DHO (trough  $\sim$  84 hours after dosing) criteria, also described in the Guidelines for Individual Dose Adjustment.

Dosing will continue up to 12 months in the absence of unacceptable toxicity or disease progression, or may be discontinued with Sponsor consent after completing at least 6 weeks of dosing.

#### **B.** Study Population

Up to 27 subjects 18 years or older with relapsed/refractory AML by World Health Organization (WHO) classification who have exhausted available therapy and who meet all inclusion/exclusion criteria will be enrolled at 3-6 sites in the United States.

#### C. Sample Size Predictions

Formal sample size calculations are not applicable to this phase 1b/2a doseadjustment and expansion study.

#### V. **General Analytical Considerations**

All analyses of safety and anti-leukemic activity for this open-label, early-phase study will be descriptive in nature and presented by dose group and overall, as appropriate, for dose-adjustment and expansion phases.

Effective Date: 13-Apr-2015 Document Number: FORM 694.01 DCN # 1372  Statistical code and outputs for analyses will be generated using SAS/STAT and SAS/GRAPH software, version 9.3 or higher, of the SAS system for Windows. Copyright © [2011] SAS Institute Inc. SAS and all other SAS Institute Inc. product or service names are registered trademarks or trademarks of SAS Institute Inc., Cary, NC, USA.

#### A. Data Sources

The study center staff will record completion and results of required study procedures in an electronic case report form (eCRF). The following external data obtained from third-party vendors for this study will be combined with eCRF data for analysis:

| Vendor<br>Name | Contact<br>Information | Data Type | Schedule | Reconciliation Items |
|---|---|---|---|---|
| Pyxant | TBD | DHO | 2 transfers during | Header data (subject |
| | | plasma | study | ID, initials, visit, lab |
| | | levels and | | date, lab time) |
| | | brequinar | | |
| | | PK results | | |

#### **B.** Multiple Study Centers

Data analyses will be pooled and not controlled for center effect.

#### C. Definition of Baseline

Baseline will be defined as the last measurement collected before the first dose of study drug. As such, height and body surface area assessed at Screening, and predose assessments made on Cycle 1 Week 1 Day 1 for weight, vital signs, hematology/chemistry, and 12-lead ECG will serve as valid baseline measures. A missing value at Cycle 1 Week 1 Day 1 will default to the Screening measurement.

For this study, since there is no day 0, the day immediately prior to study day 1 will be Day -1 [calculated as Event Date – Date of First Treatment]. For events on or after first dose of study drug, study day will be calculated as [Event Date – Date of First Treatment + 1]. Thus, first day of study drug dose will be Day 1.

#### D. Missing Data

Unless stated otherwise in sections below, missing data will not be replaced with imputed values.

#### E. Analysis Populations

Four analysis population sets will be defined for use with various analyses, namely:

Document Number: FORM 694.01
DCN # 1372
Document Title: Statistical Analysis Plan Template
Effective Date: 13-Apr-2015
Page **5** of **23** 

- The Enrolled Analysis Set will include all subjects who sign informed consent, meet the inclusion/exclusion criteria and are enrolled in the study. Demographics and disposition summaries will be reported for this set of subjects.
- The Safety Analysis Set will include all subjects who are enrolled in the study and receive at least one dose of brequinar. Subjects in this set will be used for all safety/tolerability summary tables.
- The Efficacy Analysis Set will be a subset of the Safety population with measurable AML disease at baseline and at least one post-baseline disease response assessment. Subjects in this set will be used for all efficacy summary tables.
- Pharmacokinetic Analysis Set will be a subset of the Safety population with at least 1 quantifiable plasma concentration collected post-dose without important protocol deviations/violations or events thought to significantly affect the PK. Summary tables for PK concentrations and parameters will be based on this set of subjects.

#### F. Data Display Characteristics

Data displays produced for this study will include three types—data listings, summary tables, and figures.

Unless stated otherwise, data listings will be produced for all recorded data. Data listings will simply list the data recorded on the CRF or derived for each subject. They will be ordered by treatment, subject number, and date and time of assessment, where applicable. When expedient, additional levels of ordering hierarchy may reflect subsets of assessments within subject. Additional listings may be produced for outcome measures that involve extensive procedure to derive analyzed outcomes.

Summary tables will display summary statistics calculated for each of the treatment groups, and overall. When the evolution of statistics over time is of interest, a group of rows that represent a cohort would generally be ordered chronologically.

The summary statistics displayed will be a function of the type of data associated with the summarized assessment. Continuous data will be summarized with the number of nonmissing values, mean, standard deviation (SD), minimum, median, and maximum. Categorical data will be summarized with the number of nonmissing values. Corresponding percentages will be calculated using the relevant analysis population set as the denominator, unless stated otherwise. Some continuous variables may also be grouped into categorical levels and evaluated in frequency tables.

Effective Date: 13-Apr-2015 Document Number: FORM 694.01 DCN # 1372  PK concentrations and parameters will be summarized using n (for available data), mean, SD, coefficient of variation percent (CV%), median, minimum, and maximum values. Geometric means and geometric CV% will also be calculated for PK parameters.

All PK concentrations will be reported and analyzed with the same precision as the source data provided by the bio-analytical laboratory regardless of how many significant figures or decimals the data carry.

Extra measurements (such as unscheduled or repeat assessments) will be included in subject listings but not in summary tables.

Figures will be produced as specified in sections to follow.

#### VI. **Subject Accountability**

#### A. Analysis Populations

A summary table will present counts and percent of subjects in the study analysis populations of Enrolled, Safety, Efficacy, and PK Analysis sets by treatment group.

## **B.** Disposition

All subjects who discontinue treatment or withdraw early from the study will be included in a listing. Disposition summaries will present number of subjects enrolled, number treated, and among those treated number who completed and discontinued treatment. Primary reason for discontinuation of treatment, including any of the following, will be summarized:

- Adverse event
- Physician/Sponsor decision
- Pregnancy
- Protocol defined disease progression
- Study terminated by sponsor
- Subject non-compliance/Protocol violation(s)
- Withdrawal of consent.

Counts and percentages of subjects who withdraw early from the study for any of the above reasons will also be calculated using all members of the relevant population in the relevant treatment group for the denominator.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372 

#### C. Subject Characteristics

The following subject characteristics collected for the Enrolled Analysis Set will be presented in data listings and summarized by treatment regimen and overall:

#### Demography:

- Age: Age will be calculated as the number of years elapsed between birth date and the date of the screening visit, adjusted for whether the birthday has passed as of the day of the screening visit.
- Sex at birth
- Ethnicity
- Race

#### Medical History:

- Medical history: As noted on the Medical History eCRF, any significant medical conditions present prior to signing consent will be presented in a listing and summary table. Verbatim terms will be coded using the MedDRA version 21.1 and ordered by system organ class (SOC) and preferred term (PT). At each level of summation (SOC, PT), subjects reporting more than one medical condition will be counted only once.
- AML disease information: Disease characteristics of initial diagnosis of AML recorded on the eCRF, along with time since initial diagnosis (calculated as date of informed consent – date of initial diagnosis of AML/365.25), will be listed and summarized.
- AML supplemental tests: Cytogenetics and molecular data information recorded on the eCRF will be listed, including information on karyotypic, Fluorescence in situ hybridization (FISH), and gene fusion analysis, as well as all present mutations.
- Prior cancer drug treatment: A listing will display all entries for prior cancer medications received by a subject, ordered by "Start date". A summary table will summarize the following characteristics:
  - Number of subjects reporting at least one prior cancer drug treatment.
  - Drug treatment type (Chemotherapy, Targeted therapy, Immunological, Not Applicable).
  - Drug treatment combined with radiotherapy (No/Yes).
  - Number of cycles received.
  - Best response under treatment (Complete remission, Complete remission with incomplete hematologic recovery, Complete remission with partial hematologic recovery, Morphologic

Effective Date: 13-Apr-2015 Document Number: FORM 694.01 DCN # 1372  Clear Creek Bio, Inc. / Protocol: CCB-01 IQVIA Biotech (Confidential) Project # YYA36071

> leukemia-free state, Partial remission, Stable disease, Progressive disease, Unknown).

- Relapse (derived as 'Yes' if date of relapse is not blank. 'No' otherwise).
- Prior cancer non-drug treatment: All non-drug treatments received will be listed in order of "Start date". Summary statistics will be provided for:
  - Number of subjects reporting at least one prior cancer non-drug treatment.
  - Treatment type (Radiation, Surgery, Other).
  - Intention (Palliative, Therapeutic).
  - Best response under treatment (Complete remission, Complete remission with incomplete hematologic recovery, Complete remission with partial hematologic recovery. Morphologic leukemia-free state, Partial remission, Stable disease, Progressive disease, Not applicable, Unknown).
  - Relapse (derived as 'Yes' if date of relapse is not blank. 'No' otherwise).

#### **D.** Protocol Deviations

A listing will be provided for all protocol deviations.

## VII. Safety Analyses

To meet the primary objective of the study, all safety analyses will be performed on the Safety Analysis Set of subjects.

#### A. Exposure

For each subject, the assigned dose level of brequinar (mg/m<sup>2</sup>), the assigned dose (mg), dose day, date and time taken, whether entire dose was taken, number of capsules taken, total dose taken (mg), and the reason for missed dose (partial or complete) will be listed by treatment group and visit cycle.

Summary statistics will be presented for assigned dose level, cumulative assigned dose, cumulative actual exposure (mg), total duration of treatment (calculated as the number of weeks from date of first drug dose to date of last drug dose), dose intensity (calculated as cumulative actual exposure divided by treatment duration, mg/week), relative dose intensity (calculated as a percent of cumulative actual drug dose divided by cumulative assigned dose), and any reason for missed dose.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372 

#### **B.** DHO Plasma Levels

In addition to safety/tolerability, intra-subject dosing for this study will be guided by DHO levels measured using a validated assay. A subject listing will include baseline and trough DHO levels (ng/ml), as well as the following additional characteristics noted at each scheduled visit:

- Previous assigned dose (mg/m<sup>2</sup>).
- DHO dose adjustment (dose not changed, escalated by 150 mg/m<sup>2</sup>, held, Cohort 1 dose escalation not permitted).
- Assigned dose based on DHO (mg/m<sup>2</sup>).
- PI evaluation of whether subject has acceptable safety, safety dose adjustment, and assigned dose.
- Actual dose (mg).
- Agreement between PI assessment and actual dose (No/Yes, reason for disagreement).

The above dose-modification characteristics will also be summarized by treatment group and overall.

### C. Dose Limiting Toxicities

AEs identified as protocol-defined DLTs will be listed and will include start and end dates, CTCAE grade, relationship to study drug, outcome, and action taken. Number and percentage of subjects reporting DLTs in each treatment group, and overall, will be summarized.

#### **D.** Adverse Events

AEs will be collected from time of informed consent through at least 14 days after the final dose of study medication. Any pre-existing condition that changes in severity after dosing or abnormal laboratory finding will be recorded as an AE. Events that occur prior to dosing will be recorded as medical history. A TEAE for this study will be defined as an AE occurring after the first dose of the study treatment through 30 days after the last dose of study treatment.

Verbatim terms on the eCRF will be coded using the MedDRA version 21.1 and displayed hierarchically by system organ class and preferred term. Multiple incidences of the same AE for a subject will be counted only once at the maximum CTCAE grade.

All AEs (whether TEAEs or not) will be listed by treatment group and individual subject, and include start and end dates, if the event was serious, seriousness criteria, CTCAE grade, relationship to study drug, action taken with study drug, and any other action. All TEAEs, Serious TEAEs, TEAEs that lead to study drug being permanently discontinued, and TEAEs resulting in death will be listed separately.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372  All AEs (whether TEAEs or not) will be summarized by system organ class and preferred term for each treatment group.

An overall summary table for TEAEs, and TEAEs occurring 10% or higher in the study population by preferred term and CTCAE grade will be provided. All TEAEs, grade 3 or greater TEAEs, TEAEs related to study drug (i.e., relationship to study drug deemed by the principal investigator as "Definite", "Probable", or "Possible"), grade 3 or greater TEAEs related to study drug, serious TEAEs, TEAEs leading to study drug being permanently discontinued, and TEAEs resulting in death will each be summarized by system organ class and preferred term. At each level of summation of system organ class and preferred term, subjects reporting more than one AE will only be counted once.

#### E. Deaths

All deaths and the primary cause of death will be listed.

#### F. Clinical Laboratory Results

Clinical laboratory tests for safety will be performed according to the study schedule, samples analyzed at local laboratories, and data entered directly into the electronic data capture system by site users.

Results for hematology and chemistry panels will be presented in separate data listings along with a flag for normal, abnormal not clinically significant, or abnormal clinically significant values. Listings will also be provided for pregnancy test, flow cytometry, and chromosomal/mutation testing.

Beginning with the baseline results, summaries of actual values at each assessment time point, and change from baseline will be presented by dose level and overall for each hematology and chemistry parameter. Change from baseline will be calculated as the post-baseline measurement minus the baseline measurement. If either the baseline or post-baseline value is missing, the observation will not be included in the change from baseline summary.

For hematology parameters leukocytes, hemoglobin, and platelets that can be graded using the NCI CTCAE criteria, shift tables that summarize counts and percentages of subjects by severity grade at baseline and worst post-baseline result will also be constructed.

The percentage of blasts in bone marrow ascertained via aspiration and biopsy will be listed and summarized.

#### G. Vital Signs

At designated visits, vital signs will be recorded and will include weight, temperature, heart rate, respiratory rate, and systolic and diastolic blood pressure. A listing of all vital signs, along with height and derived body surface area, will be provided. Additionally, data will be summarized by dose group and overall, using descriptive statistics at baseline, each study evaluation, and change from baseline to evaluation. Change from baseline will be calculated as the postbaseline measurement minus the baseline measurement. If either value is missing, the observation will not be included in the change from baseline summary.

#### H. 12-Lead Electrocardiogram

12-lead ECG data, obtained at scheduled visits, will be listed. Counts and percentages of subjects with normal, abnormal clinically significant, and abnormal not clinically significant evaluations will be summarized at each time point.

#### T. **ECOG Performance Status**

ECOG performance status assessed at Screening will be listed and summarized for each numeric grade.

#### J. **Physical Examination**

Confirmation of a physical examination, including date of assessment, will be listed for each scheduled time point.

#### **K.** Concomitant Medications

Any medication or treatment taken within two weeks prior to study entry as well as during the course of the study will be recorded in the eCRF. Indication for use, start date (if known), dose frequency, route, and whether ongoing or stopped will also be noted.

Verbatim terms from the eCRF will be mapped to Anatomical/Therapeutic Chemical class and Generic drug names using the WHODD version September 2018 Enhanced B2.

For each dose cohort, a listing will display all entries for medications received by a subject, ordered by "Start date". The listing will display the recorded term from the eCRF and, adjacent to that, the WHO Drug pharmacological subgroup and the anatomical main class that appears in the tables.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372  A summary table will be constructed to display the anatomical main class (1st level) of each coded medication and, within that, the pharmacological subgroup (3<sup>rd</sup> level). It will include counts and percentages of subjects who reported using at least one medication in each pharmacological subgroup.

#### L. Blood Transfusions

Any blood transfusions received up to eight weeks prior to Cycle 1 Day 1 (baseline event), and during the study, including start and end dates, blood product, total number of units received, and reason for transfusion will be listed and summarized.

## VIII. Efficacy Analyses

The secondary objectives of the study will be addressed using the Efficacy Analysis Set of subjects.

#### A. Disease Response

As per criteria defined in the ELN Guidelines by Dohner et al, 2017, disease response will be assessed at screening and post-screening visits and included in a data listing. Additionally, anti-leukemic activity will be evaluated as per the following outcomes:

Response Rates: The distribution of best overall response (BOR) of CR, CRi, CRh, MLFS, or PR will be summarized by treatment cohort and overall. Point estimates with two-sided exact 95% and 90% confidence intervals (CIs) will be included for:

- Overall response rate (ORR) defined as the proportion of subjects who achieve a best overall response of CR, CRi, CRh, MLFS, or PR.
- Complete remission rate defined as the proportion of subjects who achieve a best overall response of CR.
- Complete remission with incomplete hematologic recovery rate defined as the proportion of subjects who achieve a best overall response of CRi.
- Complete remission with partial hematological recovery rate defined as the proportion subjects who achieve a best overall response of CRh.
- Morphological leukemia-free state rate defined as the proportion of subjects who achieve a best overall response of MLFS.
- Partial remission rate defined as the proportion of subjects who achieve best overall response of PR.

Additional information on precise definitions of these response categories can be found in Section 10.3 of the protocol.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372  Duration of Response: Duration of response will be defined as the time from the first occurrence of a qualifying response of CR, CRi, CRh, MLFS, or PR, to the date when progressive disease is objectively documented or death due to any cause, whichever occurs earlier. Following the qualifying response, subjects who are alive without disease progression will be right-censored at the date of last disease evaluation. A Kaplan-Meier graph will be plotted by treatment group and estimates of median duration with associated 95% CIs will be reported.

Event-free Survival (EFS): Event-free survival will be determined from the first dose of brequinar to the date of relapse (> 5% bone marrow blasts, reappearance of blasts in blood, or development of extramedullary disease), disease progression, or death, whichever occurs first. Subjects who do not experience any of the three events will be right-censored at the latter date of disease evaluation or bone marrow sampling. A Kaplan-Meier graph will be plotted for time to the composite outcome by treatment group, and the estimate of medial survival time with 95% CI will be summarized.

Overall Survival (OS): Overall survival will be calculated as the time from the first dose of study drug to the date of death or right-censoring at the date of last subject contact. Median time to OS, with 95% CI, will be summarized and displayed graphically by treatment group using the Kaplan-Meier method.

#### **B.** Clinical Benefit

In addition to ORR, this study will examine clinical benefit to subjects. By treatment group, a summary table will report counts and percent of transfusion-dependent subjects at baseline who, in the absence of progression, CR or PR, and independent of marrow response, achieve one of the following:

- Erythroid response: Transfusion Independence (TI) for 8 or more weeks for subjects requiring at least 4 units of packed red blood cell transfusions in the previous 8 weeks. Only red blood cell transfusions given based on physician's judgment for a pretreatment hemoglobin (Hgb) of < 8.5 g/dL will count in the red blood cell TI response evaluation.
- Platelet response: TI for subjects requiring a minimum of 4 platelet transfusions in the previous 8 weeks.

#### IX. **Pharmacokinetic Analyses**

The plasma PK of brequinar and DHO will be characterized using noncompartmental analysis. Where possible, the following standard PK parameters will be calculated:

AUC<sub>0-last</sub>: Area under plasma concentration-time curve from time 0 to time of last measurable concentration.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372  Clear Creek Bio, Inc. / Protocol: CCB-01 IQVIA Biotech (Confidential) Project # YYA36071

- AUC<sub>0-inf</sub>: Area under plasma concentration-time curve from 0 to infinity.
- C<sub>max</sub>: Maximum observed plasma concentration.
- C<sub>ss</sub>: Observed plasma concentration at steady-state.
- CL: Systemic clearance.
- T<sub>max</sub>: Time to maximum plasma concentration.
- $T_{1/2}$ : Elimination half-life
- V<sub>ss</sub>: Volume of distribution at steady state.

Listings of PK concentration and parameters will be generated using the Pharmacokinetic Analysis Set of subjects. Concentration and PK parameters will also be tabulated and summarized by treatment group at baseline and scheduled time points using descriptive statistics.

A listing of derived time interval between Brequinar dosing and pre-dose PK sampling will be provided.

Mean concentration-time profiles by treatment group, as well as by-subject plots for observed concentrations of brequinar and DHO levels will be presented on linear and semi-logarithmic scales.

Relationship between PK parameters, DHO levels, and clinical outcomes (e.g. efficacy, toxicity) may be explored.

## X. Exploratory Analyses

This study will endeavor to explore the following aims:

Relationship between DHODH inhibition and the efficacy and safety of brequinar:

Identify molecular and cellular biomarkers predictive of antitumor level and/or treatment resistance including cytogenetics, molecular profiling and flow cytometry during and after treatment:

Evaluate global gene expression profiles, DNA methylation profiles, and other potential prognostic markers as predictors of antitumor activity and/or resistance to treatment.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372 Document Title: Statistical Analysis Plan Template Page **15** of **23** 

#### **Changes from Analyses Planned in Protocol** XI.

There are no significant changes to the analyses planned in the study protocol.

Effective Date: 13-Apr-2015 Page **16** of **23** Document Number: FORM 694.01 DCN # 1372

## XII. References

- 1. CCB-01 Protocol\_ver\_5\_16OCT2018-FINAL.pdf
- 2. CCB-01 Protocol ver6 30APR2019 FINAL signed 15MAY2019.pdf
- 3. Dohner H, Estey E, Grimwade D, Amadori S, Applebaum FR, Buchner T, et al. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood 2017; 129(4); 424-447.

Document Number: FORM 694.01 Effective Date: 13-Apr-2015 DCN # 1372 